CLINICAL TRIAL: NCT01322464
Title: A Phase I Study to Assess the Effect of Food on the Single-Dose Bioavailability of Sativex, and to Compare the Single and Multiple Dose Pharmacokinetics of Sativex at Three Dose Levels
Brief Title: Study to Assess Food Effect on Sativex Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GWCP0601
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Food Effect
Keywords: Sativex; bio-availability; cannabinoid; pharmacokinetics
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 Fasted-Fed (Experimental): 4 sprays Sativex in fasted state, followed by wash-out followed by 4 sprays Sativex in fed state.
  Followed by 4 sprays daily in fasted state.
  Interventions: Drug: Sativex
- Group 1 Fed-Fasted (Experimental): 4 sprays sativex in fed state followed by wash-out followed by 4 sprays Sativex in fasted state.
  Followed by 4 sprays daily in fasted state.
  Interventions: Drug: Sativex
- Group 2 (Experimental): 2 sprays Sativex daily in fasted state.
  Interventions: Drug: Sativex
- Group 3 (Experimental): 8 sprays sativex daily in fasted state.
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — 4 sprays Sativex in fasted state on Day 1. 4 sprays Sativex in fed state on Day 4. 4 sprays Sativex daily in fasted state Days 5-13.
  Arms: Group 1 Fasted-Fed
Drug: Sativex — 4 sprays Sativex in fed state on Day 1. 4 sprays Sativex in fasted state on Day 4. 4 sprays Sativex daily in fasted state Days 5-13.
  Arms: Group 1 Fed-Fasted
Drug: Sativex — 2 sprays Sativex daily in fasted state Days 4-13.
  Arms: Group 2
Drug: Sativex — 8 sprays Sativex daily in fasted state Days 4-13.
  Arms: Group 3

SUMMARY:
Study to assess effect of food on the bioavailability of a single dose of Sativex and to measure its' pharmacokinetics after a single and multiple doses.

DETAILED DESCRIPTION:
This was an open-label, randomised, ascending dose, 2-way crossover food-effect study incorporating a parallel single and multiple dose components in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 45 years of age (inclusive).
* Body mass index to be between 18 to 30 kg/m2 (inclusive) as calculated by weight(Kg)/height(m2).
* Subjects were to have no clinically significant abnormal findings on physical examination, ECG, medical history, or clinical laboratory results during screening.
* Subjects were to, in the opinion of the investigator, have no clinically significant abnormal findings of renal and hepatic function as determined by serum creatinine, total bilirubin, and transaminase levels.
* Subjects were to be non-users of tobacco products (minimum of 6 months prior to the start of the study).
* Subjects were to have a negative screen for HIV I and II, HBsAg, and antibody to Hepatitis C virus.
* Subjects were to have a negative urine screen for alcohol, drugs of abuse (screening only), and cotinine.
* Subjects were to use an appropriate barrier method of contraception (condom and spermicide) in addition to having their female partner use another form of barrier contraception (e.g.female condom or occlusive cap with spermicide) during the study and for 3 months following administration of the study drug.
* Subjects were able to comply with the protocol and the restrictions and assessments therein.
* Subjects were to give voluntary written informed consent to participate in the trial.

Exclusion Criteria:

* Subjects were not to have a history or presence of significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* Subjects were not to have any history or presence or family history of schizophrenia, other psychotic illness, severe personality disorder, depression, or other significant psychiatric disorder.
* Subjects were not to have a postural drop of 20 mmHg or more in systolic blood pressure at screening.
* Subjects were not to have participated in a previous clinical trial within 90 days prior to study initiation.
* Subjects were not to have donated plasma within 90 days prior to study initiation.
* Subjects were not to have donated blood within 90 days prior to study initiation.
* Subjects were not to have had an abnormal diet or substantial changes in eating habits within 30 days prior to study initiation.
* Subjects were not to have had treatment with any known enzyme-altering agents (barbiturates, phenothiazines, cimetidine etc.) within 30 days prior to or during the study.
* Subjects were to have no history of known hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
* Subjects were not to use any prescription medication within 14 days prior to or during the study.
* Subjects were not to use any over-the-counter medication within 7 days prior to or during the study.
* Subjects were not to have a history of alcohol or drug abuse within 2 years prior to the study (subjects with a history of previous use of cannabis were not excluded unless they had used cannabis or cannabinoid based medicine within 30 days prior to study drug administration or were unwilling to abstain for the duration of the study).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Primary PK Endpoints
  Cmax, AUC(0-inf), T-half and CL/F: under fasting conditions (Group 1, Day 1 and 4 fasted data) and under fed conditions (Group 1 Day 1 and 4 fed data)

SECONDARY OUTCOMES:
Secondary PK measures
  Cmax, Tmax, AUC(0-t), t-half, CL/F, Varea/F from Day 4 (Groups 2 and 3) and from fasted subjects on days 1 and 4 (Group 1) Cmax, Cmin, Tmax, AUC(0-t), Flux from Day 12 data (all groups)
Safety and tolerability of Sativex

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's Drug Research Unit, Quintiles Ltd., London, United Kingdom

REFERENCES:
- [Result] Stott CG, White L, Wright S, Wilbraham D, Guy GW. A phase I study to assess the effect of food on the single dose bioavailability of the THC/CBD oromucosal spray. Eur J Clin Pharmacol. 2013 Apr;69(4):825-34. doi: 10.1007/s00228-012-1393-4. Epub 2012 Oct 4. PMID 23052407
- [Result] Stott CG, White L, Wright S, Wilbraham D, Guy GW. A phase I study to assess the single and multiple dose pharmacokinetics of THC/CBD oromucosal spray. Eur J Clin Pharmacol. 2013 May;69(5):1135-47. doi: 10.1007/s00228-012-1441-0. Epub 2012 Nov 22. PMID 23179176